CLINICAL TRIAL: NCT04681950
Title: Assessment of Unsupervised Self-Collected Saliva Sample Compared to Clinician CollectedSaliva Sample and Clinician Collected Anterior Nares Sample in a COVID-19 and Influenza A/Influenza B Screening Program
Brief Title: Assessment of Self-Collected Sample Compared to Clinician Collected Sample in COVID-19 and Influenza Program
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Biocerna LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 00047586
Record Dates: First submitted 2020-12-22; First posted 2020-12-23 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Subjects Possibly Exposed to COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We are trying to see whether a self-collected saliva swab in the home setting is as good as or better than a study clinician-collected anterior nose swab in evaluating whether you are positive for COVID-19 or Influenza A/Influenza B. You may have no symptoms, so you may be positive and capable of spreading the infection to others and you don't know it. Knowing whether you are positive is important because you would have to quarantine and not go out to prevent spreading the infection to others.

DETAILED DESCRIPTION:
In some research studies, saliva has been shown to be as good as or even better than an anterior nares or nasopharyngeal specimen in detecting SARS-CoV-2; we are interested in making sure that is the case. Being able to collect a specimen at home and mail it in would help with patient compliance and would reduce the need for clinicians (nurses or other health care professionals) to use personal protective equipment (PPE), which is in short supply. Also, people would not have to go to a healthcare facility or other testing site to have the COVID-19 or the Influenza A/Influenza B testing done. We are using a sensitive method (RT-PCR) to look for the three viruses.

Once you have had the anterior nose swab collected by the study clinician, your participation would last only as long as it takes to complete the self-collected saliva collection and return the sample to the researchers. The self-collection of the saliva specimen should be collected as soon as possible after the collection of anterior nares and saliva samples by the clinician You will mail in the saliva swab in a prepaid mailer no later than 10 days after sample collection and the result will be available within one day of our lab receiving the swab. Once our lab receives your specimen, the gift card which you received will be activated and your participation will be complete. Biocerna, LLC (Fulton, Maryland), is the commercial laboratory to which the research subjects' samples will be shipped and tested.

We anticipate approximately 500 subjects will be enrolled. You qualify because you live in a location which is reporting an increased number of COVID-19 positive cases. Incidence of Influenza A/Influenza B is also useful to track to find out whether social distancing and/or wearing masks decreases the number of Influenza A/Influenza B cases during the winter months.

ELIGIBILITY:
Inclusion Criteria: Patients will qualify because they live in a location which is reporting an increased number of COVID-19 positive cases. Incidence of Influenza A/Influenza B is also useful to track to find out whether social distancing and/or wearing masks decreases the number of Influenza A/Influenza B cases during the winter months.

-

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We anticipate approximately 500 subjects will be enrolled. You qualify because you live in a location which is reporting an increased number of COVID-19 positive cases. Incidence of Influenza A/Influenza B is also useful to track to find out whether social distancing and/or wearing masks decreases the number of Influenza A/Influenza B cases during the winter months.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Matching results from different collection types | 3 days from the time of collection
  Samples will be collected by the patient and a HCP

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sanders, Principal Investigator — Vice President of Clinical Operations
Locations (1):
- Biocerna LLC, Fulton, Maryland, United States